CLINICAL TRIAL: NCT01452373
Title: DHEA + Acolbifene Against Vasomotor Symptoms (Hot Flushes) in Postmenopausal Women (Placebo Controlled, Double Blind and Randomized Phase III Study to Evaluate the Effects of 12-Week Treatment With DHEA (Prasterone) and Acolbifene on Vasomotor Symptoms (Hot Flushes) in Postmenopausal Women)
Brief Title: Dehydroepiandrosterone (DHEA) + Acolbifene Against Vasomotor Symptoms (Hot Flushes) in Postmenopausal Women
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EndoCeutics Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: ERC-207
Record Dates: First submitted 2011-10-12; First posted 2011-10-14 (Estimated); Last update posted 2013-12-11 (Estimated); Status verified 2013-12

CONDITIONS: Vasomotor Symptoms; Hot Flushes
Keywords: Hot flush(es); Hot flash(es); Vasomotor symptoms; Dehydroepiandrosterone (DHEA); Prasterone; Acolbifene; Selective estrogen receptor modulator (SERM); Antiestrogen; Menopause; Postmenopausal women
MeSH Terms: conditions — Hot Flashes | interventions — Dehydroepiandrosterone; ritetronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Control (placebo) (Placebo Comparator)
  Interventions: Drug: Placebo
- DHEA + Acolbifene (Experimental)
  Interventions: Drug: DHEA and Acolbifene

INTERVENTIONS:
Drug: Placebo — Placebo DHEA capsules (2) + placebo acolbifene capsule (1); daily oral dosing for 12 weeks.
  Arms: Control (placebo)
Drug: DHEA and Acolbifene — DHEA capsules (2 x 50 mg) + acolbifene capsule (1 x 20 mg); daily oral dosing for 12 weeks.
  Other Names: Prasterone; dehydroepiandrosterone; EM-652.HCl
  Arms: DHEA + Acolbifene

SUMMARY:
The purpose of this Phase III trial is to evaluate the efficacy of oral administration of dehydroepiandrosterone (DHEA) combined with acolbifene (a selective estrogen receptor modulator (SERM)) on vasomotor symptoms (hot flushes) in postmenopausal women.

ELIGIBILITY:
Main Inclusion Criteria:

* Postmenopausal women (non-hysterectomized or hysterectomized).
* Women between 40 and 75 years of age.
* Willing to participate in the study and sign an informed consent.
* Women having many moderate to severe hot flushes.
* For non-hysterectomized women, willing to have an endometrial biopsy at baseline and end of-study.

Main Exclusion Criteria:

* Undiagnosed abnormal genital bleeding.
* Hypertension equal to or above 140/90 mm Hg.
* The administration of any investigational drug within 30 days of screening visit.
* Endometrial hyperplasia (simple or complex hyperplasia with or without atypia), cancer or endometrial histology showing proliferative, secretory or menstrual type characteristics at histologic evaluation of endometrial biopsy performed at screening.

Ages: 40 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 238 (Actual)
Dates: Start 2011-10; Primary Completion 2012-12 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Co-primary endpoint: change from baseline to week 12 in frequency of moderate to severe hot flushes. | 12 weeks
Co-primary endpoint: change from baseline to week 12 in severity of moderate to severe hot flushes. | 12 weeks

SECONDARY OUTCOMES:
Change from baseline to week 12 on vaginal atrophy parameters (superficial cells, parabasal cells, pH, vaginal atrophy symptoms). | 12 weeks
Change from baseline to week 12 on sexual function and quality of life as evaluated by appropriate questionnaires. | 12 weeks
Tolerance to systemic administration of DHEA and acolbifene. | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Leonello Cusan, M.D., Ph.D., Principal Investigator — Clinique de Recherche en Traitements Hormonaux, 2785 blvd Laurier - Suite SS5, Quebec, QC, Canada
Locations (15):
- Canada (15):
  - EndoCeutics site # 06, Bathurst, New Brunswick
  - EndoCeutics site # 70, Burlington, Ontario
  - EndoCeutics site # 69, Corunna, Ontario
  - EndoCeutics site # 73, Kitchener, Ontario
  - EndoCeutics site # 71, London, Ontario
  - EndoCeutics site # 72, Newmarket, Ontario
  - EndoCeutics site # 68, Sarnia, Ontario
  - EndoCeutics site # 04, Drummondville, Quebec
  - EndoCeutics site # 12, Montreal, Quebec
  - EndoCeutics site # 02, Québec, Quebec
  - EndoCeutics site # 01, Québec, Quebec
  - EndoCeutics site # 18, Saint Romuald, Quebec
  - EndoCeutics site # 08, Shawinigan, Quebec
  - EndoCeutics site # 11, Sherbrooke, Quebec
  - EndoCeutics site # 67, Victoriaville, Quebec

REFERENCES:
- [Background] Labrie F. Drug insight: breast cancer prevention and tissue-targeted hormone replacement therapy. Nat Clin Pract Endocrinol Metab. 2007 Aug;3(8):584-93. doi: 10.1038/ncpendmet0559. PMID 17643129
- [Background] Labrie F. DHEA, important source of sex steroids in men and even more in women. Prog Brain Res. 2010;182:97-148. doi: 10.1016/S0079-6123(10)82004-7. PMID 20541662
- [Background] Labrie F, Belanger A, Labrie C, Candas B, Cusan L, Gomez JL. Bioavailability and metabolism of oral and percutaneous dehydroepiandrosterone in postmenopausal women. J Steroid Biochem Mol Biol. 2007 Oct;107(1-2):57-69. doi: 10.1016/j.jsbmb.2007.02.007. Epub 2007 Jun 8. PMID 17627814
- [Background] Labrie F, Champagne P, Labrie C, Roy J, Laverdiere J, Provencher L, Potvin M, Drolet Y, Pollak M, Panasci L, L'Esperance B, Dufresne J, Latreille J, Robert J, Samson B, Jolivet J, Yelle L, Cusan L, Diamond P, Candas B. Activity and safety of the antiestrogen EM-800, the orally active precursor of acolbifene, in tamoxifen-resistant breast cancer. J Clin Oncol. 2004 Mar 1;22(5):864-71. doi: 10.1200/JCO.2004.05.122. PMID 14990642
- [Background] Labrie F, Labrie C, Belanger A, Simard J, Gauthier S, Luu-The V, Merand Y, Giguere V, Candas B, Luo S, Martel C, Singh SM, Fournier M, Coquet A, Richard V, Charbonneau R, Charpenet G, Tremblay A, Tremblay G, Cusan L, Veilleux R. EM-652 (SCH 57068), a third generation SERM acting as pure antiestrogen in the mammary gland and endometrium. J Steroid Biochem Mol Biol. 1999 Apr-Jun;69(1-6):51-84. doi: 10.1016/s0960-0760(99)00065-5. PMID 10418981